CLINICAL TRIAL: NCT05589142
Title: Effect of Early Time Restricted Eating and BCAA Supplementation vs. Early Time Restricted Eating Alone on Body Composition
Brief Title: Effect of Early Eating and BCAA Supplementation on Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Dr. Peter Lemon, Western University, Canada
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121699
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: eTRE (Early Time Restricted Eating) With BCAA; eTRE (Early Time Restricted Eating)
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTRE with BCAA (Experimental): participants allocated to this group will only consume calories during 0800h and 1600h daily. Prior to sleep, participants will consume a single bolus of 5.6g of BCAA.
  Interventions: Behavioral: Time Restricted Eating
- eTRE (Active Comparator): participants allocated to this group will only consume calories during 0800h and 1600h daily.
  Interventions: Behavioral: Time Restricted Eating

INTERVENTIONS:
Behavioral: Time Restricted Eating — Eating calories only during a specific feeding window.

SUMMARY:
To our knowledge, as of this day there are only four studies which examined the effects of eTRE with a duration of 12 weeks. There are no studies that examined this phenomenon beyond 12 weeks, one study that lasted five weeks and four studies that lasted 4 weeks or less, some even days. The four studies that lasted 12 weeks in duration all have opportunities to improve upon, which will be discussed here. The first study performed by Gabel et al., focused primarily on measuring body weight, not body composition in older adults. The eating window also began later in the morning at 1000h and finished at 1800h. There also was no restriction on participants consuming caffeine during the fasting window. The second study conducted by Gasmi et al., was focused on strictly older male participants that were active and healthy, again, without measuring body composition. The third study conducted by Wilkinson et al., did not measure body composition and the eating window lasted 10 hours instead of 8. The fourth study performed by Chow et al., examined eTRE with adults aged 45+/-12 years old and did not mention any exclusion criteria based upon physical activity levels or restrictions on caffeine/artificial sweetener intake during the fasting window. Furthermore, none of the studies mentioned above examined eTRE against eTRE with BCAA supplementation directly. We believe that the proposed study will address the concerns mentioned previously and further knowledge associated with eTRE.

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of early with BCAA supplementation (5.6g) and early time restricted eating alone on body composition in overweight and obese young adults. It is hypothesized that early time restricted eating with BCAA will provide a more desirable effect (lower fat mass and greater lean mass) on body composition for the participants.

The sample will include 28 overweight/obese young adults, male and female, ranging in age from 18-39 that volunteer to participate in the study. This sample size is justified assuming a standard deviation of 1.5 based on previous studies and using a power of 80% with the statistical significance of 0.05 the resulting n would be 2(1.5)^2*(0.84+1.96)^2/5=7 (Kadam, P., & Bhalerao, S. (2010). Sample size calculation. International journal of Ayurveda research, 1(1), 55). To account for dropouts/non-interest in participation, 14 matched participants will be recruited for each group. All individuals must give written informed consent in order to participate in the study. Exclusion criteria include self-reported: diabetes, smoking, CVD, pregnancy, weight loss medication, physical activity level greater than low/sedentary (7500 steps daily), unstable weight (>4kg loss/gain) for 3 months prior to study commencement.

All participants will be required to have their Body Composition measured using non-invasive densitometry (BodPod). The procedure poses no risk to the participant and takes approximately 5 minutes to complete. This procedure will take place initially one week prior to study commencement and then every 4 weeks after study commencement until the 12 weeks of the study duration are complete. This results in a total of 4 measurements. Upper body strength measurements will be recorded one week prior to commencement of the study and once again after study completion using a 3-rep maximal bench press test. Lower body strength measurements will be recorded one week prior to commencement of the study and once again after study completion using a 3-rep maximal leg press test. Completion of a health-related quality of life questionnaire one week prior to commencement of the study and once again after study completion is also required.

One week prior to study commencement participants will come to the Exercise Nutrition Research Laboratory and initial body composition will be recorded along with baseline upper body strength, lower body strength and health-related quality of life scores. Once the study has commenced, participants will adhere to the daily time windows depending on which group they are randomly assigned. The early time restricted eating with BCAA (5.6g) group will begin their food intake at 0800 h and finish at 1600 h. The early time restricted eating group alone will begin their caloric intake at 0800 h and finish at 1600 h. During the fasting window participants are encouraged to drink plenty of fluids (ad libitum) BUT they must not contain calories, artificial sweeteners or caffeine. Participants will also notify Reed Zehr through email of adherence to their timing windows on a weekly basis. Body composition measurements will take place every 4 weeks upon study commencement. Upon completion of the study, participants will return to the Exercise Nutrition Research Laboratory and final measurements will be recorded of body composition, upper body strength, lower body strength, and health-related quality of life using the same procedure initially.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25
* 18-39 yo
* <7500 steps daily

Exclusion Criteria:

* diabetes, smoking, CVD (self-reported)
* BMI < 24.9
* pregnant, medication for weight loss (self-reported)

  -> 7500 steps/day
* employed in shift work position
* unstable weight for 3 months prior to study (>4kg weight loss/gain)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
body composition | <5 mins
  fat mass vs fat-free mass

SECONDARY OUTCOMES:
upper body strength | < 15 mins
  3 rep max, bench press
lower body strength | <15 mins
  3 rep max, leg press
subjective quality of life questionnaire | < 5 mins
  4 question survey

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No